CLINICAL TRIAL: NCT06150612
Title: Unwinding Anxiety for Migraine: Pilot
Acronym: UAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeshiva University (Other)
Responsible Party: Principal Investigator, Elizabeth Seng, Associate Professor, Yeshiva University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20216986
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Migraine; Anxiousness
MeSH Terms: conditions — Migraine Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unwinding Anxiety (Experimental)
  Interventions: Behavioral: Unwinding Anxiety

INTERVENTIONS:
Behavioral: Unwinding Anxiety — In the Unwinding Anxiety arm, participants will receive 6 weeks of an educational app and weekly facilitated mindfulness groups.

SUMMARY:
This is a pilot study that aims to understand the feasibility and acceptability of a mobile health educational app plus group-based mindfulness therapy on anxiety and migraine-related disability among people with migraine.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Meets diagnostic criteria for migraine
* Reports anxiety symptoms of 5 or more on GAD-7
* Has a smartphone

Exclusion Criteria:

* Under the age of 18
* Presence of suicidal ideation
* Reports severe depression on PHQ-9
* Lack of group readiness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-03 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 weeks
  Average number of facilitated mindfulness group sessions attended out of 6 weekly sessions

SECONDARY OUTCOMES:
Acceptability | Assessed at 6 weeks, immediately post-intervention
  Average Credibility Score from the Credibility/Expectancy Questionnaire [min = 3; max = 27; higher scores indicate higher credibility]

OTHER OUTCOMES:
Change in Anxiety | Change from Week 0 to Week 10
  Patient Reported Measurement Outcome System - Anxiety Short Form Score [min = 37; Max = 83; higher scores indicate higher levels of anxiety symptoms]
Change in Headache-Related Disability | Change from Week 0 to Week 10
  Headache Disability Inventory Score [min = 0; max = 100; higher scores indicate higher levels of headache-related disability]

CONTACTS AND LOCATIONS:
Locations (1):
- Rousso Building, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to investigators with an approved IRB and DUA.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be made available 12 months after primary study completion.
Access Criteria: Contact investigators.